CLINICAL TRIAL: NCT06146673
Title: A Multidimensional Study of Premenstrual Syndrome, Body Image, Physical Activity and Sleep Quality Among Women in Reproductive Age
Brief Title: A Multidimensional Study of Premenstrual Syndrome and Body Image
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Dózsa-Juhász Olívia, Subject Teacher, University of Pecs
Other Study IDs: BM/23899-1/2023
Record Dates: First submitted 2023-11-17; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Body Image; Premenstrual Syndrome; Sleep; Physical Inactivity
Keywords: physical activity; premenstrual syndrome; body mass index; 24 hour movement behaviour; sleep quality; body image
MeSH Terms: conditions — Premenstrual Syndrome; Sedentary Behavior; Motor Activity; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this cross-sectional study is to investigate the influencing factors of body image in women of reproductive age. The main question[s] it aims to answer are:

* Is there a connection between physical activity, body mass index and body image?
* Is there a connection between body image, premenstrual syndrome and sleep quality? Participants will fill out a complex online questionnaire.

DETAILED DESCRIPTION:
During the research, the researchers use a quantitative method, in which the participants fill out the Knowledge of the Female Body Scale, the Global Physical Activity Questionnaire, the Body Appreciation Scale, the Sleep Quality Scale and the Premenstrual Assessment Form Short Form, as well as a general health status questionnaire. and a self-made questionnaire containing socio-demographic questions. In the course of the research, we form a sub-sample, on which we carry out further instrumental tests to monitor body composition and physical activity. The number of participants is approx. There will be 500 women between the ages of 18 and 45, who will be selected through targeted sampling. During the research, the data are processed in the SPSS v28.0 program and the following statistical methods are used: Kolmogorov-Smirnov and Shapiro-Wilk normality tests, Spearman and Pearson correlation analysis, Pearson chi-square test, linear regression analysis. During the research, the safety of the participants and the ethical rules are strictly observed.

ELIGIBILITY:
Inclusion Criteria:

* women
* between the ages of 18-45 years
* regular menstruation

Exclusion Criteria:

* older than 45 years
* pregnancy
* amenorrhoea
* premature ovarian failure

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women between the ages of 18-45 who reported symptoms of PMS during the period of parameterization of the target group
Sampling Method: Non-Probability Sample
Enrollment: 329 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Body Image | 1 day
  points; Body Appreciation Scale (13 item version, 4 subscales); 1-5 point scale, minimum score: 13 points; maximum score: 65 points, the higher the points the worse the body image

SECONDARY OUTCOMES:
Global Physical Activity Questionnaire | 1 week
  MET/min 16 questions Assessing work-, travel-related and recreational physical activity and the hours spent sitting.
Sleep Quality | 1 day
  points; Sleep Quality Scale (28 items, 6 subscales); 0-3 point scale, minimum score: 0 points; maximum score: 84 points, the higher the points the worse the sleep quality
Premenstrual syndrome | 1 day
  points; Premenstrual Assessment Form Short Form Questionnaire (10 item version); 1-6 point scale, minimum score: 10 points; maximum score: 60 points, the higher the points the worse the symptoms
Body mass index | 1 day
  kg/m^2
Knowledge of he Female Body | 1 day
  points; Knowledge of the Female Body Scale 26 questions 0-17=low knowledge 18-26=high knowledge
Health Literacy | 1 day
  points; Brief Health Literacy Screening Tool (4 questions) 1-5 point scale, minimum score: 4 points; maximum score: 20 points, 4-12 points=inadequate 13-16=marginal 17-20=adequate

CONTACTS AND LOCATIONS:
Overall Officials: Olívia Dózsa-Juhász, BSc, Study Chair — University of Pecs
Locations (1):
- University of Pécs, Pécs, Baranya, Hungary

REFERENCES:
- [Derived] Premusz V, Kovacs KA, Skriba E, Tandor Z, Szmatona G, Dozsa-Juhasz O. Socio-Economic and Health Literacy Inequalities as Determinants of Women's Knowledge about Their Reproductive System: A Cross-Sectional Study. Epidemiologia (Basel). 2024 Sep 26;5(4):627-642. doi: 10.3390/epidemiologia5040044. PMID 39449387